CLINICAL TRIAL: NCT04235491
Title: Longitudinal Coverage With Evidence Development Study on Micra AV Leadless Pacemakers
Brief Title: Longitudinal Coverage With Evidence Development Study on Micra AV Leadless Pacemakers (Micra AV CED)
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Micra AV CED Study
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Micra AV leadless pacemaker therapy: All Medicare patients implanted with a Micra AV leadless pacemaker system
- Dual Chamber Transvenous pacemaker: All Medicare patients implanted with full system (e.g. lead and generator) dual-chamber transvenous pacemakers

SUMMARY:
The primary purpose of the study is to meet the CMS mandated Coverage with Evidence Development requirement in the National Coverage Determination for Leadless Pacemakers as they apply to Medtronic Micra devices. The study uses administrative claims data of the Medicare population implanted with Micra AV leadless pacemakers or dual-chamber transvenous pacemakers. Patients are enrolled through submission of claims or encounter data to CMS.

DETAILED DESCRIPTION:
The Micra AV CED study is a study of the Medicare beneficiary population implanted with Micra AV leadless pacemakers or dual-chamber transvenous pacemakers and will be executed by analyzing administrative claims data. The study consists of two primary objectives: estimate the (1) acute overall complication rate, and (2) the 2-year survival rate of patients implanted with a Micra AV leadless pacemaker. As part of the secondary objectives of the study, a comparative analysis of Micra AV leadless pacemakers to dual-chamber transvenous pacemakers will be conducted.

The analysis will be in CMS claims data and is subject to a central IRB. However, individual hospitals are not engaged in research and local IRB oversight is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries implanted with a Micra AV leadless pacemaker (CPT 0387T or 33274 or ICD-10 PCS 02HK3NZ) on or after the study start date will be included in the study.

or

- Medicare beneficiaries implanted with a dual-chamber ventricular transvenous pacemaker [CPT 33208 or 33213 or 33214 or ICD-10 PCS ((0JH606Z or 0JH636Z) + (02H60JZ or 02H63JZ or 02H70JZ or 02H73JZ) + (02HK0JZ or 02HK3JZ))] on or after the study start date.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will include all Medicare patients with continuous claims data implanted with a Micra AV leadless pacemaker or a full-system dual-chamber transvenous pacemaker in any US location.
Sampling Method: Probability Sample
Enrollment: 37000 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Acute complication rate | 30 days
  Micra AV leadless pacemaker system and/or procedure related complications at 30 days. Acute complications include embolism/thrombosis, event at the puncture site, cardiac effusion/perforation, device-related complication, or other complications following the implantation of a Micra AV leadless pacemaker system. Subjects' administrative claims data will be reviewed to determine the occurrence of an acute complication.
The 2-year survival of patients implanted with a Micra AV leadless pacemaker | 2 years
  Estimate the 2-year survival rate of patients implanted with a Micra AV leadless pacemaker

SECONDARY OUTCOMES:
Chronic complication rate | 6 months
  Chronic complications are a subset of acute complications that may also occur within six months following the implantation of a Micra AV leadless pacemaker. Micra AV leadless pacemaker system and/or procedure related complications at six months. Subjects' administrative claims data will be reviewed to determine the occurrence of a chronic complication.
Device-related re-intervention rates | 2 years
  Device-related re-interventions are procedures associated with the insertion/replacement, revision, or removal or either a leadless or transvenous pacemaker system or components following the index implantation of a Micra AV leadless pacemaker. Device-related re-intervention rates will be reported at six month intervals for two years following the index implantation of a single-chamber ventricular pacemaker. Subjects' administrative claims data will be reviewed to determine the occurrence of a device-related re-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael El Chami, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Chami MF, Higuera L, Longacre C, Stromberg K, Crossley G, Piccini JP. Two-year outcomes of Micra AV leadless pacemakers in the Micra AV CED study. Europace. 2024 Nov 1;26(11):euae273. doi: 10.1093/europace/euae273. PMID 39485833